CLINICAL TRIAL: NCT01710267
Title: Rivaroxaban Laboratory Monitoring in Switzerland 2: Therapeutic Dose (RivaMoS 2)
Acronym: RivaMoS2
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Dr. med. Walter A. Wuillemin, MD, PhD (Other)
Collaborators: Research Foundation, Division of Hematology, Luzerner Kantonsspital, Switzerland (Unknown); Bayer (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Dr. med. Walter A. Wuillemin, MD, PhD, Chief, Division of Hematology and Central Hematology Laboratory, Luzerner Kantonsspital, Switzerland, Luzerner Kantonsspital
Organization: Luzerner Kantonsspital (Other)
Other Study IDs: 12041
Record Dates: First submitted 2012-10-17; First posted 2012-10-19 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2015-03

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for coagulation assays
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observation group: This group includes all volunteers of this observation study.

SUMMARY:
Rivaroxaban (RXA; brand name Xarelto®) is an oral direct factor Xa inhibitor that is applied for prophylaxis of venous thromboembolism after major orthopedic surgery. Additionally, RXA is approved by Swissmedic to be used at a therapeutic dose for primary therapy of VTE and for prophylaxis of cerebrovascular events in non-valvular atrial fibrillation.

This is an explorative laboratory study to evaluate the intra-individual variability of RXA conc. in time and to standardize assays among 9 Swiss laboratories to determine RXA conc.

DETAILED DESCRIPTION:
Rivaroxaban (RXA; brand name Xarelto®) is an oral direct factor Xa inhibitor that is applied for prophylaxis of venous thromboembolism (VTE) after major orthopedic surgery of the lower limbs such as hip and knee replacement surgery. Additionally, RXA is approved by Swissmedic to be used at a therapeutic dose for primary therapy of VTE and for prophylaxis of cerebrovascular events in non-valvular atrial fibrillation.

Monitoring of RXA concentration (conc.) is generally not required because of its stable pharmacokinetic and pharmacodynamic profile, even in patients with renal insufficiency. However, there are several clinical situations, in which it may be desirable to measure the RXA plasma conc. The range of RXA conc. is wide among individuals with typical peak levels of median 244 µg/L (IQR 175-360) and trough levels of median 32 µg/L (IQR 19-60) with once daily doses of 20 mg RXA.

This is an explorative laboratory study to evaluate the intra-individual variability of RXA conc. in time and to standardize assays among 9 Swiss laboratories to determine RXA conc.

ELIGIBILITY:
Inclusion Criteria:

Male, aged 18-65 years

* No known comorbidity or disease
* No known galactose intolerance, lactase deficiency or glucose galactose malabsorption
* Taking no other medicaments
* No history for disorders regarding hemostasis
* Initial screening laboratory test showing normal values for liver/pancreas function (ALAT,ASAT,gGT, alkalic phosphatase, bilirubin, amylase, lipase), kidney function (creatinine), hematogram (white blood cell count, hemoglobin, platelet count), and coagulation parameters ("Gerinnungsstatus" with PT, aPTT, fibrinogen, thrombin time)
* written informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy male volunteers aged 18-65 years
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of RXA on trough and peak RXA conc. values in time | 14 days

SECONDARY OUTCOMES:
Evaluation of the effect of RXA on coagulation assays in time | 14 days
  coagulation assays such as PT, PTT, individual coagulation factors, PiCT, ROTEM, multiplate

CONTACTS AND LOCATIONS:
Overall Officials: Walter A Wuillemin, MD PhD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Kantonsspital, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Derived] Studt JD, Alberio L, Angelillo-Scherrer A, Asmis LM, Fontana P, Korte W, Mendez A, Schmid P, Stricker H, Tsakiris DA, Wuillemin WA, Nagler M. Accuracy and consistency of anti-Xa activity measurement for determination of rivaroxaban plasma levels. J Thromb Haemost. 2017 Aug;15(8):1576-1583. doi: 10.1111/jth.13747. Epub 2017 Jul 17. PMID 28574652
- [Derived] Fontana P, Alberio L, Angelillo-Scherrer A, Asmis LM, Korte W, Mendez A, Schmid P, Stricker H, Studt JD, Tsakiris DA, Wuillemin WA, Nagler M. Impact of rivaroxaban on point-of-care assays. Thromb Res. 2017 May;153:65-70. doi: 10.1016/j.thromres.2017.03.019. Epub 2017 Mar 21. PMID 28343143
- See also: Division of Hematology and Central Hematology Laboratory, Luzerner Kantonsspital, Switzerland — https://www.luks.ch/standorte/luzern/kliniken/medizin/haematologie.html